CLINICAL TRIAL: NCT03665844
Title: Smart Sleep In-home Validation Extension Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SRC-AI-SMILES-2018-10210
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Healthy; Sleep Deprivation; Insufficient Sleep Syndrome
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: 1 week baseline, 3 weeks active condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SmartSleep Boost Off (Placebo Comparator): Participants wear the device for baseline data collection in boost off mode. There is no intervention. This is known as SmartSleep Boost Off mode.
  Interventions: Device: SmartSleep Boost Off
- SmartSleep Boost On (Active Comparator): Participants wear the device for 3 weeks in boost on mode. This is known as SmartSleep Boost On mode.
  Interventions: Device: SmartSleep Boost On

INTERVENTIONS:
Device: SmartSleep Boost On — SmartSleep device can be configured to two different settings. SmartSleep Boost On setting provides soft audio tones during the night.
  It's a non-invasive portable light weight device designed to stimulate deep slow wave sleep (SWS).
  Arms: SmartSleep Boost On
Device: SmartSleep Boost Off — SmartSleep device can be configured to two different settings. SmartSleep Boost Off provides no audio tones.
  Arms: SmartSleep Boost Off

SUMMARY:
This study is a nonrandomized, unblinded, uncontrolled case series clinical trial validating the SmartSleep product, including SleepMapper app in the home setting. It is intended to provide data related to product use and cognitive testing incorporating a longer baseline period for comparison purposes. It will include adults (21-50 yr. old) who are working full time and report shortened sleep due to lifestyle. For the purposes of this study, shortened sleep is defined as sleeping at least 5 hrs. of sleep per night, and sleeping less than or equal to 7 hrs. at least 3 nights per week. Participants also increase their sleep duration by ≥ 1 hour on the weekends. In addition, participants report a sleep latency ≤ 30 minutes less than or equal to 3 nights per week. Participants are generally healthy individuals who have not been diagnosed with any sleep-related medical conditions. In addition, participants diagnosed with major organ system diseases or requiring oxygen therapy are excluded from participation. Up to 75 individuals will be consented in order to complete a total of 50 participants using a nonrandomized design. The study involves an initial screening visit followed by home use of the SmartSleep device with SleepMapper app. The home use will include an initial week of baseline use followed by 3 weeks of use with boost on. Study staff will contact participants after the first week of use as a reminder. Participants will be asked to complete a battery of cognitive tests upon wake up each morning. Participants will be asked to complete a question twice daily during the home use period. Additional phone calls may occur on an as needed basis if issues arise. The final visit will be an in facility visit in which all study equipment will be returned. The anticipated study duration will be up to 6 weeks (including the 4 weeks of use period).

DETAILED DESCRIPTION:
Study procedures

Visit 1 (Screening) Procedures (up to 2 hours):

Participants will be asked to report to the research site for a daytime visit. A detailed interview will be performed verifying eligibility criteria, as well as a review of work and non-work schedules. After a full explanation of the protocol and after all the participants' questions have been answered, they will be asked to sign the consent form.

Participants will complete the following baseline information:

Demographics Questionnaires Medical History Questionnaire Review of Current Medications Height, Weight, Head Measurements Cognitive Assessment training

Once eligibility confirmed, participants will be trained in the use of the SmartSleep device, including pairing and syncing of the SleepMapper app

Home Use (weeks 1-4) All participants will be asked to wear the device consecutively every night. The anticipated study participation is expected to be one month of use (+ 2 weeks based on participant schedule). All participants will wear the device for 1 week of baseline use. Post one week of use (+/- 2 days), participants will the active mode. Participants will continue nightly home use of the SmartSleep with boost enabled for the next 3 weeks.

Participants will be asked to complete the cognitive testing daily after wake up. Cognitive tests should be performed at the same time each morning following the same routine.

Participants will be asked to complete the a question twice daily.

During the study if a participant's medical history or medication changes, they will be asked to inform the study team. Participants will be asked during the course of the study if they experience any discomfort, red marks, etc.

Study completion (final visit) Participants will be asked to return to the lab for a final study visit. They will be asked to bring their study materials.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Live in the US
* Able to read, write and speak English
* Adult volunteers aged 21-50
* Smartphone owner (iOS 9+ or Android 5.0+ OS)
* Access to home Wi-Fi for syncing of SmartSleep data and cognitive testing
* Working full time schedule [Note: Full time is considered a 32 hour work week start time at 7am or later]
* Suffer from short sleep due to lifestyle

  * Gets less than 7 hours of sleep at least 3 days a week (via self-report)
  * Get at least 5 hours of sleep per night 7 nights a week (via self-report)
  * Gets 1 extra hour of sleep on the weekends (via self-report of extended nightly sleep or daytime nap)

Exclusion Criteria:

* Individuals who self-report severe contact dermatitis or an allergy to silver
* Diagnosed as having any of the following conditions (via self-report):

  * Sleep Apnea
  * Insomnia
  * Restless legs syndrome
  * Parasomnia
  * Epilepsy/Seizures
* Diagnosed as having any major organ system disease such as congestive heart failure, neuromuscular disease, renal failure, cancer, chronic obstructive pulmonary disease, respiratory failure or respiratory insufficiency, or patients requiring oxygen therapy (via self-report)
* High Risk of Obstructive Sleep Apnea (OSA) based on Questionnaire
* Daily caffeine intake > 650 mg
* History of moderate hearing loss (via self-report)
* Currently working night shift or rotating shift
* Head circumference <54 cm (21 in) or >66 cm (26 in)
* Individuals who self-report taking longer than 30 minutes more than 3 times a week to fall asleep once they turn lights off
* Individuals who self-report regularly taking sleeping pills (more than once per week), including prescription or over the counter (OTC) pills such as Ambien, Tylenol PM or Zzzquil
* Pregnant (via self-report)
* Employee of Philips or spouse of a Philips employee
* Employee (or spouse of an employee) of a company that designs, sells, or manufactures sleep-related products
* Not able to comply with study procedures

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
The effects of the auditory stimulation delivered by the SmartSleep device in adults with shortened sleep schedules due to lifestyle as determined by changes in the cumulative (CSWA) or average slow-wave activity. | 4 weeks
  Efficacy will be evaluated based on the average of seven nights of use collecting baseline data compared to the average of twenty one nights of active SmartSleep, while in the home setting. SWA accumulation over Non-Rapid Eye Movement (NREM) sleep (CSWA) will be analyzed for each night in the active condition using as reference the average CSWA across baseline nights.

SECONDARY OUTCOMES:
Change in performance of the Matrix reasoning task (MRT) correlated to the changes in CSWA over the trial period. | 4 weeks
  Performance of the MRT during baseline and active use weeks of the SmartSleep Device will be compared to changes in CSWA over the trial period.
Change in performance of the Digital Symbol Substitution Task (DSST) correlated to the changes in CSWA over the trial period. | 4 weeks
  Performance of the DSST during baseline and active use weeks of the SmartSleep Device will be compared to changes in CSWA over the trial period.
Change in performance of the Psychomotor Vigilance Testing -Brief (PVT) correlated to the changes in CSWA over the trial period. | 4 weeks
  Performance of the PVT during baseline and active use weeks of the SmartSleep Device will be compared to changes in CSWA over the trial period.
Change in sleepiness/alertness as measured by a 7 point scale correlated to the changes in CSWA over the trial period. | 4 weeks
  Change in sleepiness/alertness as measured by a 7 point scale during baseline and active use weeks of the SmartSleep Device will be compared to changes in CSWA over the trial period.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Lung & Sleep Associates, Lehigh Acres, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No. This data will remain with Florida Lung & Sleep Associates and Philips